CLINICAL TRIAL: NCT05642338
Title: A Multicenter Prospective Cohort Study Comparing Random Biopsies Versus Wide-Area Transepithelial Brush-Sampling (WATS) for Surveillance of Barrett's Esophagus, the WATS-EURO2 Study
Acronym: WATSEURO2
Status: Recruiting | Type: Observational
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, Jacques J.G.H.M. Bergman, prof.dr., Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Other Study IDs: NL81868.018.22
Record Dates: First submitted 2022-11-28; First posted 2022-12-08 (Actual); Last update posted 2022-12-08 (Actual); Status verified 2022-12

CONDITIONS: Barrett Esophagus; Esophageal Adenocarcinoma; Diagnosis
Keywords: detection; Barrett Esophagus; WATS3D; forceps Biopsies; Dysplasia
MeSH Terms: conditions — Barrett Esophagus; Adenocarcinoma Of Esophagus; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — samples of the distal barrett mucosa in the oesophagus collected with forceps biopsies and the WATS3D brush
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (2):
- cohort 1 dysplastic cohort: 208 BE patients referred for work up after diagnosis of LGD, HGD or earlystage cancer in the last 18 months.
  Interventions: Diagnostic Test: WATS3D
- Cohort 2: non-dysplastic cohort: 208 patients under standard BE surveillance without a diagnosis of dysplasia in last 18 months.
  Interventions: Diagnostic Test: WATS3D

INTERVENTIONS:
Diagnostic Test: WATS3D — the WATS3D brush samples the esophagus by abresing the tissue. the brush is directed through the workingchanel of endoscope into the oesophagus
  Other Names: CDxx WATS3D brush

SUMMARY:
The investigators aim to study the rate of developing a biopsy-based diagnosis of high-grade dysplasia (HGD) and EAC in BE patients in a prospective cohort of 208 BE patients at high risk of progression (i.e. after endoscopic removal of visible lesions containing HGD/EAC and/or a diagnosis of low-grade dysplasia (LGD)) as well as in 208 BE patients with a nondysplastic BE (NDBE) undergoing standard BE surveillance. In these patients the investigators will combine biopsy sampling with WATS at baseline and all follow-up endoscopies during a 3- year follow-up period. This will allow us to study the natural history of WATS-positive-biopsynegative- cases and of WATS-specific outcomes such as basal-crypt dysplasia. The study also allows us to collect specimens for future biomarker studies that may help to predict progression to HGD/EAC in the absence of morphological features of dysplasia.

DETAILED DESCRIPTION:
Esophageal adenocarcinoma (EAC) is a disease with a poor prognosis at advanced stages.

Identifying esophageal adenocarcinoma at an early stage allows for endoscopic treatment to reduce mortality and morbidity for these treated patients. Adequate surveillance strategies with appropriate risk stratification are therefore essential. The current endoscopic surveillance protocol relies on systemic four-quadrant biopsy at 2-cm intervals of the BE segment, with additional targeted biopsies from visible abnormalities.

Obtaining random biopsies is time consuming, and it results at best in sampling less than 5% of the BE surface area . Thus, significant sampling error is inevitable. Sampling the BE segment with a brush has the theoretical advantage of larger field sampling and might therefore increase the detection of dysplasia. Conventional brush cytology samples however, suffer from superficial sampling and difficult analysis of the thick tissue smear by a twodimensional cytology microscope. The WATS system (developed by CDx Diagnostics) consists of a trans-epithelial cytology brush designed to sample cells from all three layers of the epithelium and the diagnosis of the brush specimen by advanced computer image analysis system at CDx Diagnostics.

These advantages over conventional cytology may make this system an important diagnostic tool in BE surveillance . In the European WATS study ("Euro-WATS1") the WATS-system was compared with random biopsies in a cohort of patients referred with low-grade dysplasia (LGD), high-grade dysplasia (HGD) or early cancer after removal of all visible abnormalities. Eligible cases underwent random biopsies and WATS brushings after randomizing the order of sampling.

The study showed no significant differences in the detection rate for HGD or EAC between random biopsies and WATS brushings. The brush detected 39/48 HGD/EAC cases versus 30/48 for random biopsies (p=0.12). The value of the WATS-3D brush as an adjunct to random forceps biopsies however, was 48/147 vs 30/147; difference 12%, with a number needed to treat of 8. Moreover, the brush had a significantly shorter procedure time than random biopsies with a larger difference in longer BE segments. Another strength of the WATS brush, compared to random biopsies, is that it paves the way towards a preferred (future) trans-oral sampling instead of endoscopic sampling. Key element in the adjunctive value of WATS is the clinical relevance of "WATS-positive-biopsy-negative". One may argue that the morphological changes of dysplasia-positive WATS samples clearly correspond to those defining dysplasia in biopsy samples and therefore are merely different representations of the same disease which is now diagnosed at an earlier stage. Others argue that the WATS-system, by being more sensitive to detect dysplasia, simply dilutes the disease reservoir with clinically less severe cases which do not warrant the same therapeutic approach as in cases with a biopsy based diagnosis of dysplasia. The natural history of "WATS-positive-biopsy-negative" cases can, however, not be investigated in the EUROWATS1 study because this was a transversal study with no subsequent follow-up and with the vast majority of cases having undergone ablation therapy based on their referral diagnosis and/or outcome of the endoscopic resection of visible lesions. Another limitation of the EURO-WATS1 study was the relatively high rate of WATS brushings that were deemed ineligible for assessment of the smears. In the study 23/172 (13%) of cases had suboptimal WATS samples, despite the fact that the corresponding cellblocks showed adequate cellularity. It appears that the logistics in the endoscopy suite and/or storage of samples prior to transportation and evaluation at CDx may have had flaws. Therefore, a second European WATS study ("WATS EURO 2 study") will be performed in which, after the baseline endoscopy with WATS brushing and random biopsies, endoscopic follow-up is continued until a biopsy-based diagnosis of HGD or cancer is made. The WATS EURO 2 study will therefore allow us to study the natural history of WATS-positive-biopsynegative cases, will enable us to re-evaluate the role of the WATS-3D brush as a potential substitute for random sampling, after optimizing sample collection and preparation in the study. Finally, the samples collected in this study will also allow us to perform future biomarker studies on both the brush and biopsy material, to find the best sampling method for biomarker risk stratification in the future. It is undisputed that patients referred with LGD, HGD or early cancer should have all visible lesions removed by ER techniques. In general, the endoscopic resection specimen will then show a diagnosis of HGD or early cancer. Follow-up studies have shown that the chance of the development of metachronous HGD/EAC in the remaining BE segment is about 10% per year. Therefore ablation therapy is advised for the remaining BE segment.

The same 10% annual progression rate to HGD/EAC applies for patients with a confirmed diagnosis of LGD. For these patients, guidelines suggest that ablation therapy may be a valid alternative to subsequent surveillance. The actual decision to ablate the remaining Barrett's segment after endoscopic resection of HGD/EAC or to prophylactically ablate for LGD, is made on a per patient basis in which age and comorbidity are important additional factors to be taken into account. Follow-up studies after ER of visible lesions containing HGD/EAC have found that metachronous lesions are all found at an endoscopically treatable stage with the majority of patients not developing recurrent disease. The same holds for prophylactic ablation in cases with LGD: a significant proportion of patients will not progress or not even manifest their baseline diagnosis of LGD upon follow-up. In the SURF-study, 30% of the LGD-patients randomized to endoscopic surveillance did not have their LGD diagnosis reproduced during 4 subsequent endoscopies in 3-years follow-up and all cases that progressed to HGD/EAC were diagnosed at an endoscopically curable stage. Furthermore, RFA still is accompanied by complications such as esophageal stenosis and requires multiple hospital visits. Even upon complete endoscopic eradication of all Barrett's mucosa, guidelines still dictate endoscopic surveillance after ablation virtually at the same frequency as for Barrett's cases not prophylactically treated. Therefore, keeping Barrett's patients under strict endoscopic surveillance after ER of visible lesions or for flat LGD is an acceptable strategy that does not divert from current guidelines.

In the current study, the investigators aim to study the rate of developing a biopsy-based diagnosis of HGD/EAC in Barrett's patients at high risk of progression (i.e. after endoscopic removal of visible lesions containing HGD/EAC and/or a diagnosis of LGD) as well as in patients in a standard Barrett's surveillance program. In these patients the investigators will combine biopsy sampling with WATS brushing at baseline and all follow-up endoscopies. This will allow us to study the natural history of WATS-positive-biopsy negative case and of WATS-specific outcomes such as basal-crypt dysplasia, and to further evaluate the role of the WATS brush as a potential substitute to random biopsies.

The study also allows us to collect specimens for future biomarker studies that may help to predict progression to HGD/EAC in the absence of morphological features of dysplasia.

ELIGIBILITY:
Inclusion Criteria:

* Patients age: ≥ 18 years
* BE with a circumferential extent of ≥2cm and a total maximum extent of ≤18cm (in case of prior ER: BE length is measured after ER). Or a circumferential extent of 0-1 cm with a maximum extent of ≥4cm.
* Cohort 1: Patients referred for work-up of IND, LGD, HGD or low-risk cancer (m1 to sm1, without lympho-vascular invasion and poor differentiation), either diagnosed in random biopsies or in prior endoscopic resection specimen within 18 months prior to baseline endoscopy
* Cohort 2: Patients with known BE without a diagnosis of dysplasia in the last 18 months, enrolled in endoscopic surveillance programs
* Ability to give written, informed consent and understand the responsibilities of participation

Exclusion Criteria:

* Patients with visible lesions according to the Paris classification at the time of the WATS and random biopsy testing (prior endoscopic resection is allowed)
* Patients with high-risk cancer after endoscopic resection: either sm2/3 invasion, poor differentiation, lympho-vascular invasion, or R1 vertical resection margin
* Patients within six weeks after endoscopy with biopsies and/or ER
* History of esophageal or gastric surgery other than Nissen fundoplication
* History of esophageal ablation therapy
* Presence of esophageal varices
* Subject has a known history of unresolved drug or alcohol dependency that would limit ability to comprehend or follow instructions related to informed consent, post-treatment instructions, or follow-up guidelines

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Barrett Esophagus patient enrolled in a surveillance cohort
Sampling Method: Probability Sample
Enrollment: 416 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2027-05-01 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
HGD/EAC | 3 years after last inclusion
  The concordance/discordance for the diagnosis HGD/EAC between random biopsies and WATS brushings collected at the baseline endoscopy and follow-up endoscopies.

SECONDARY OUTCOMES:
The proportion of patients diagnosed with HGD/EAC on endoscopic biopsies (targeted or random) or endoscopic resection specimens during a maximum follow-up of 3 years | 3 years after last inclusion
  The proportion of patients diagnosed with HGD/EAC on endoscopic biopsies (targeted or random) or endoscopic resection specimens during a maximum follow-up of 3 years
The rate of progression to HGD/EAC after a WATS-positive-biopsy-negative diagnosis for HGD/EAC | 3 years after last inclusion
  The rate of progression to HGD/EAC after a WATS-positive-biopsy-negative diagnosis for HGD/EAC

CONTACTS AND LOCATIONS:
Overall Officials: prof Bergman, MD, PhD, Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Locations (1):
- Amsterdam University Medical Centre, loc. VUmc, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No